CLINICAL TRIAL: NCT04482023
Title: Emotional Support and Stress Management Activities Offered by Nurses to Patients Diagnosed With COVID-19 During Hospital Admission
Brief Title: Emotional Support and Stress Management in Patients Diagnosed With COVID-19
Acronym: WWCOVID-19
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Corporacion Parc Tauli (Other)
Responsible Party: Principal Investigator, Montserrat Montaña, Principal Investigator, Clinical Research, Corporacion Parc Tauli
Other Study IDs: 2020663
Record Dates: First submitted 2020-07-21; First posted 2020-07-22 (Actual); Last update posted 2021-03-24 (Actual); Status verified 2021-03

CONDITIONS: COVID-19
Keywords: Nursing care; Anxiety; Loneliness; Fear; Education; COVID-19
MeSH Terms: conditions — COVID-19; Anxiety Disorders

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Nurses COVID 19: Nurses from any unit of the Consortium Parc Taulí Corporation who have been in direct care of patients diagnosed with COVID 19 between March 9, 2020 and May 15, 2020
  Interventions: Behavioral: Training video on anxiety, fear and loneliness in the COVID-19 environment.

INTERVENTIONS:
Behavioral: Training video on anxiety, fear and loneliness in the COVID-19 environment. — Video with the actions identified as essential to address the diagnosis of anxiety, fear and loneliness in the environment COVID-19 identified by a group of experts.

SUMMARY:
The aim of the study is to identify the knowledge that CCSPT nurses have in relation to care aimed at addressing anxiety, fear or loneliness and the use they have made of it in the recent crisis. The design of the research/action will also enable the training of the participating professionals to improve nursing care in these areas in the future

DETAILED DESCRIPTION:
This is a cross-sectional descriptive study with a research/action design to be carried out at the Consorci Corporació Sanitària Parc Taulí (CCSPT). The aim of this study is to identify the knowledge that CCSPT nurses have in relation to care aimed at coping with anxiety, fear or loneliness and the use that they have made of it in the recent crisis. By its design, the research/action will allow the training of these nurses to improve nursing care of these aspects in the future. This is a population-based study, in which all CCSPT nurses who have carried out care work during the COVID-19 crisis period will be invited to participate. The variables collected will be age, sex, academic level, usual work shift, care given to reduce anxiety, fear, loneliness, coping style and self-pity. Quantitative variables will be described by their mean and standard deviation, while qualitative variables will be described in absolute and relative frequencies. A linear or non-parametric correlation will be made between the score on the self-pity and coping scales and the number of actions identified and/or performed referred to by the nurses and the calculation of the Pearson or Spearman correlation coefficient, as appropriate. Comparison of the number of actions between high activity and low activity (70% cut) coping nurses using the Mann-Whitney U test

ELIGIBILITY:
Inclusion Criteria:

* Nurses from any unit of the Consortium Parc Taulí Corporation who have been in direct care of patients diagnosed with COVID 19 between March 9, 2020 and May 15, 2020

Exclusion Criteria:

-

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: CCSPT nurses
Sampling Method: Non-Probability Sample
Enrollment: 150 (Estimated)
Dates: Start 2021-03-23 (Actual); Primary Completion 2021-04-30 (Estimated); Study Completion 2021-04-30 (Estimated)

PRIMARY OUTCOMES:
Rate of care actions identified by nurses | 6 months after care
  % of care actions identified by nurses

SECONDARY OUTCOMES:
Rate of care actions taken by nurses | 6 months after care
  % of care actions taken by nurses

CONTACTS AND LOCATIONS:
Overall Officials: Montserrat Montaña, PhD, Principal Investigator — Corporación Parc Taulí
Locations (1):
- Montserrat Montaña, Sabadell, Barcelona, Spain